CLINICAL TRIAL: NCT03927040
Title: An Open-Label Extension Study Investigating the Safety and Efficacy of Transcranial Electromagnetic Treatment Against Alzheimer's Disease
Brief Title: Transcranial Electromagnetic Treatment Against Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroEM Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM1000-1
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer Disease; Alzheimer Disease, Late Onset
Keywords: Alzheimer's Disease; Transcranial Electromagnetic Treatment; Cognitive Assessment; Alzheimer's markers in blood and CSF
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TEMT Administration (Experimental): Subjects in this arm will received Transcranial Electromagnetic Treatment (TEMT) once daily for a 4-month treatment period utilizing the MemorEM 1000 head device.
  Interventions: Device: MemorEM 1000

INTERVENTIONS:
Device: MemorEM 1000 — The MemorEM 1000 device is self-contained and has been designed for in-home daily electromagnetic treatment in the radiofrequency range, allowing for complete mobility and comfort in performing daily activities during treatment. The device has a custom control panel that is powered by a rechargeable battery. This control panel/battery box is worn on the upper arm and wired to specialized emitters in the head cap worn by the subject. The device provides global treatment to forebrain. For each of the 120 days of in-home treatment, a single 1-hour treatment will be administered by the subject's caregiver, who will position the device on the patient's head and monitor treatment.

SUMMARY:
This is an extension of EM 1000-1 wherein subjects who participated in the original study have been given the opportunity to participate in a 4-month extension of TEMT. Seven of the eight subjects in the original EM 1000-1 agreed to participate in this study extension. The time between completion of the initial study's 2-month treatment period and the beginning of this extension study's 4-month treatment period will range from 4 months to 13 months (due to staggered start of treatment in the initial study). This extension study's primary objective is to determine the effects of a follow-up treatment period of 4-months on performance of Alzheimer's Disease (AD) subjects in the same comprehensive array of cognitive tasks they performed in the initial 2-month treatment study. Baseline cognitive performance will be compared to performance at both 2-months into treatment and at the end of the 4-month treatment period. Secondary objectives include analysis of blood and CSF for AD markers and evaluation of safety throughout the treatment period.

DETAILED DESCRIPTION:
The present study is an Open-Label within-patient (single arm) extension study of our Open-Label initial study (EM1000-1) whereby seven of the eight Alzheimer's subjects participating in the initial study agreed to participate. The present study is intended to continue evaluation of the safety and efficacy of Transcranial Electromagnetic Treatment (TEMT) in patients with mild-to-moderate Alzheimer's Disease who had previously participated in the initial Open-Label study. The study duration for each subject is approximately 4 1/2 months, which involves a total of four clinical visits: pre-baseline, baseline, 2-months into treatment, and at treatment completion (4-month into treatment).

This extension study will utilize the same MemorEM 1000 head devices (designated as NSR) as in the initial 2-month treatment study, but will involve daily treatment for a longer four month period. Only one 1-hour treatment will be administered per day rather than the two 1-hour treatments per day administered in the initial 2-month study because: 1) the extension study involves a longer period of treatment, and 2) preliminary results from the initial 2-month study show a strong carry-over effect of treatment on cognitive performance after the 2-month treatment period had been completed (14 days after end of treatment).

Cognitive safety/efficacy will be evaluated using the same battery of cognitive tasks as in the initial study. These include ADAS-cog (primary outcome), and secondary cognitive outcomes of Rey AVLT, MMSE, ADCS-ADL, Digit span, Trails A & B, and clock draw tasks. Additional secondary outcomes involve analysis of blood and CSF (collected at baseline, 2-months and/or 4-months into treatment) for various beta-amyloid and tau protein species. As another secondary outcome, safety of TEMT will be monitored by regular Adverse Events Assessment, physiologic monitoring, and patient daily diaries maintained by the caregiver.

Expected Results: The investigators expect that 4-months of once-daily TEMT will not present any significant sides effects or safety issues to the seven subjects who were initially provided the same treatment twice-daily for 2-months. The investigators further expect that cognitive measures will be stable and/or improve by the end of the the treatment period. In addition, changes in blood/CSF levels of various beta-amyloid and tau species are anticipated that reflect the mechanisms of TEMT action.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild or moderate stage of Alzheimer's Disease, according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* MMSE score 16 to 26
* Physical clearance for study participation as evaluated by the clinician.
* Caregiver (spouse, family member, etc.) who agrees to and is capable of taking care and being responsible for the participation of the patient in the study (keeping a diary of health measures they collect on the patient at home, logging the patient's condition daily, and assuming responsibility for administering daily in-home treatment). Caregiver to have non-impaired mental abilities and normal motor skills, as determined by the investigators at screening. The definition of caregivers for this study is adults providing unpaid care to relatives or friends to help them take care of themselves in such activities as managing finances, shopping, preparing meals, and going to doctor appointments.
* Agreement to participate in approximately 18 weeks during the study.
* Normal to near-normal vision and hearing with correction as needed (e.g. corrective lenses, hearing aid).
* Fluent in English
* Minimum of 8th grade education
* Head circumference between 53 - 60 cm (to minimize variability in head antenna locations)
* If medicated for AD, then use of cholinesterase inhibitors and/or memantine for at least 3 months, on stable dose for at least 60 days prior to screening, and maintenance on that dose for the period of this study.
* All other non-AD medications must be stable for a period of 4 weeks prior to screening

Exclusion Criteria:

* Severe agitation
* Mental retardation
* Unstable medical condition
* Use of benzodiazepines or barbiturates 2 weeks prior to screening
* Pharmacological immunosuppression
* Participation in a clinical trial with any investigational agent within 6 months prior to study enrollment and no history of immunotherapy research participation
* History of Epileptic Seizures or Epilepsy
* Patients with major depression (not controlled with medication), bipolar disorder or psychotic disorders or any other neurological or psychiatric condition (whether now or in the past). The investigator will obtain this information from available patient medical records, history provided by the patient and caregiver, interview, and neurological exam.
* Alcoholism or drug addiction as defined by DSM-IV within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
* Patients with metal implants in the head, (i.e. cochlear implants, implanted brain stimulators, aneurysm clips) with the exception of metal implants in mouth
* Patients with vitamin B12 deficiency, abnormal thyroid function, or personal history of either any clinically defined medical disorder or any clinically defined neurological/psychiatric disorder (other than AD), including (but not limited to):, stroke, brain lesions, , cerebrovascular condition, other neurodegenerative disease, significant head trauma (loss of consciousness greater than half an hour, or related anterograde amnesia), multiple sclerosis; or personal history of previous neurosurgery or brain radiation
* Patients with any signs or symptoms of increased intracranial pressure, as determined in a neurological exam.
* Patients with demonstrated brain micro-hemorrhages (more than 5) at screening
* Patients with a score of 4 or higher on the Hachinski Test
* Patients with a score of 2 or less on the Global Deterioration Scale
* Patients with CDR Global Score of 0, 0.5, or 3
* Patients with hypertension that is unresponsive to anti-hypertensive medications
* Patients with a history of migraine headaches occurring more than once a month
* Patients with a history of cancer within last 3 years (basal cell and squamous cell carcinomas will be considered on a case by case basis by investigator)
* Patients chronically taking anticoagulants or anti-platelets (at discretion of PI)
* Pregnant women and women who have the ability to become pregnant
* Patients with compressed hair thickness of more than 5mm (which could increase distance between head antennas and the scalp).
* Cardiac pacemakers
* Implanted medication pumps
* Intracardiac lines
* Significant heart disease

Ages: 63 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
ADAS-cog score | Change from baseline ADAS-cog at two and four months into treatment
  ADAS-cog is the standard/benchmark test of cognitive performance evaluated in Alzheimer's treatment-based clinical trials.

SECONDARY OUTCOMES:
Levels of Blood and CSF Alzheimer's markers | Changes from baseline at two and four months into treatment
  Blood and CSF will be analyzed for beta-amyloid and tau species
Adverse Event Assessment | Change from baseline Adverse Event Assessment at two and four months into treatment
  AEA will be the primary safety outcome measures
Rey AVLT score | Changes from baseline Rey AVLT score at two and four months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
Digit span score | Changes from baseline Digit span score at two and four months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
MMSE score | Changes from baseline MMSE score at two and four months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
Global Deterioration score | Changes from baseline GDS at two and four months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition.
Trails A & B score | Changes from baseline in Trails A & B scores at two and four months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition
Clock draw score | Changes from baseline in Block draw score at two and four months into treatment
  This is a secondary cognitive outcome to assess effects of treatment on cognition

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Smith, MD, Principal Investigator — University of South Florida Health / Byrd Alzheimer's Institute
Locations (1):
- Byrd Alzheimer's Institute, University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
It is not anticipated that IPD will be shared with other researchers.

REFERENCES:
- [Background] Arendash GW. Review of the Evidence that Transcranial Electromagnetic Treatment will be a Safe and Effective Therapeutic Against Alzheimer's Disease. J Alzheimers Dis. 2016 May 30;53(3):753-71. doi: 10.3233/JAD-160165. PMID 27258417
- [Background] Arendash GW, Mori T, Dorsey M, Gonzalez R, Tajiri N, Borlongan C. Electromagnetic treatment to old Alzheimer's mice reverses beta-amyloid deposition, modifies cerebral blood flow, and provides selected cognitive benefit. PLoS One. 2012;7(4):e35751. doi: 10.1371/journal.pone.0035751. Epub 2012 Apr 25. PMID 22558216
- [Background] Arendash GW. Transcranial electromagnetic treatment against Alzheimer's disease: why it has the potential to trump Alzheimer's disease drug development. J Alzheimers Dis. 2012;32(2):243-66. doi: 10.3233/JAD-2012-120943. PMID 22810103
- [Background] Dragicevic N, Bradshaw PC, Mamcarz M, Lin X, Wang L, Cao C, Arendash GW. Long-term electromagnetic field treatment enhances brain mitochondrial function of both Alzheimer's transgenic mice and normal mice: a mechanism for electromagnetic field-induced cognitive benefit? Neuroscience. 2011 Jun 30;185:135-49. doi: 10.1016/j.neuroscience.2011.04.012. Epub 2011 Apr 13. PMID 21514369
- [Background] Arendash GW, Sanchez-Ramos J, Mori T, Mamcarz M, Lin X, Runfeldt M, Wang L, Zhang G, Sava V, Tan J, Cao C. Electromagnetic field treatment protects against and reverses cognitive impairment in Alzheimer's disease mice. J Alzheimers Dis. 2010;19(1):191-210. doi: 10.3233/JAD-2010-1228. PMID 20061638
- [Background] Mori T, Arendash GW. Electromagnetic field treatment enhances neuronal activity: Linkage to cognitive benefit and therapeutic implications for Alzheimer's Disease. J Alzheimer's Dis and Parkinsonism 2011; 1:102, http://dx.doi.org/10.4172/2161-0460.1000102.